CLINICAL TRIAL: NCT06382233
Title: PRecocious biOmarkers oF Unilateral ureTero-pelvic jUnction obstRuction in childrEn
Brief Title: The PRO-FUTURE Project
Acronym: PRO-FUTURE
Status: Recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: University of Milan (Other); A.O.R.N. Santobono-Pausilipon (Unknown); University of Modena and Reggio Emilia (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Pierluigi Marzuillo, Associate Professor, University of Campania Luigi Vanvitelli
Other Study IDs: PRO-FUTURE project
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Ureteropelvic Junction Obstruction; Chronic Kidney Diseases
Keywords: Ureteropelvic junction obstruction; Biomarkers; Single-Cell; Extracellular vesicles; Congenital anomalies of the kidney and urinary tract
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (3mL) will be collected at the time of pre-surgical kidney function evaluation by serum creatinine measurement in both UPJO patients and controls. Spots of urines (4-5 spots with a total volume of 150-200 mL) will be collected by sterile bag or mid-stream (before sedation) and vesical catheter (during sedation) until the start of surgical intervention. Later, only for UPJO patients, urines will be collected from bladder by sterile bag or mid-stream i) after 7 days from the pyeloplasty, and ii) after 2 months and iii) after 12 months when follow-up kidney ultrasounds will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Babies with unilateral UPJO: Children aged 0-5 years with unilateral UPJO. Unilateral UPJO will be defined as an hydronephrosis needing of surgical correction on the basis of at least 2 of the following criteria: APDP ≥ 30 mm, SRF less than 40% at the Mag3S, SRF with delta > 10% at follow-up Mag3S compared with the first Mag3S, delayed wash-out following diuretic administration, progressive increase of the APDP at follow-up kidney ultrasounds, 4th degree hydronephrosis.
  Interventions: Diagnostic Test: Identification of Diagnostic Biomarkers
- Controls of babies with unilateral UPJO: Children aged 0-5 years needing of surgical correction for hernia, hydrocele, phimosis or cryptorchidism.
  Interventions: Diagnostic Test: Identification of Diagnostic Biomarkers

INTERVENTIONS:
Diagnostic Test: Identification of Diagnostic Biomarkers — Urinary single-cell and EVs screening to stage the intrarenal injury and repair processes in UPJO babies and identification of the whole blood gene expression profiling of babies with unilateral UPJO. Data deriving from patients with unilateral UPJO will be compared with data deriving from controls.

SUMMARY:
The goal of this observational study is to learn about specific biomarkers of unilateral ureteropelvic junction obstruction (UPJO) in children undergoing surgical intervention for unilateral UPJO compared with controls. The main question it aims to answer are:

* Are Urinary single-cell and extracellular vesicles (EVs) screening useful to stage the intrarenal injury and repair processes in UPJO babies?
* Do babies with unilateral UPJO have a whole blood gene expression profiling (WBGEP) allowing an accurate unilateral UPJO diagnosis?

DETAILED DESCRIPTION:
Congenital anomalies of the kidney and urinary tract (CAKUT) are the main cause of chronic kidney disease in children. UPJO is the most common CAKUT. It is defined as impeded urine outflow from the renal pelvis to the ureter, which may result in progressive kidney damage (KD). Renal imaging is the current diagnostic approach, even if substantial shortcomings are present to reliably determine a significant obstruction. Consequently, a follow up is often needed with the risk of progressive KD. The main hypothesis of this proposal is that biofluids (whole blood and urine) could allow a more precise diagnosis and risk stratification of unilateral UPJO compared with the available diagnostic techniques.

In this project the investigators define the UPJO as an hydronephrosis needing of surgical correction according to 2 of the following criteria: anterior-posterior diameter of the pelvis (APDP) ≥ 30 mm, split renal function (SRF) < 40% at the Tc99mMag3 scintigraphy (Mag3S), SRF with delta > 10% at follow-up Mag3S, delayed wash-out, progressive increase of the APDP at follow-up ultrasounds, and 4th degree hydronephrosis.

The investigators will extensively investigate for specific biomarkers of UPJO at different levels. The investigators will focus 1. on the urine by investigating for intrarenal remodeling processes and searching for kidney-specific biomarkers by urinary single-cell and EVs screening (aim 1). Moreover, based on the hitherto revealed capability of blood cells to perceive organ-specific illnesses, 2. the investigators will perform WBGEP of babies with unilateral UPJO to identify early biomarkers of disease progression (aim 2).

For the aims 1 and 2, the investigators will enroll 85 patients aged 0-5 years, 35 with unilateral UPJO and 50 controls without hydronephrosis needing surgical correction for hernia, hydrocele or phimosis.

This project could improve the management of patients with suspect of UPJO -starting from birth- by a better understanding of the pathophysiological mechanisms underlying KD and by the identification of early biomarkers of obstruction, reducing the costs and the complications related to either a tardive or not needed surgical correction and reducing the risk of KD development.

ELIGIBILITY:
Inclusion Criteria:

* unilateral UPJO
* 0-5years of age

Exclusion Criteria:

* bilateral UPJO
* previous surgical intervention on the urinary tract
* bladder or lower urinary tract symptoms or malformations
* nephro- or urolithiasis, vesicoureteral reflux
* urinary tract infections.

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Definition of cases (patients with UPJO): in this project, the investigators define the UPJO as an hydronephrosis needing of surgical correction on the basis of at least 2 of the following criteria: APDP ≥ 30 mm, SRF less than 40% at the Mag3S, SRF with delta > 10% at follow-up Mag3S compared with the first Mag3S, delayed wash-out following diuretic administration, progressive increase of the APDP at follow-up kidney ultrasounds, 4th degree hydronephrosis. Otherwise, the hydronephrosis will be defined as non-obstructive.
  Definition of controls: babies aged 0-5 years and needing of surgical correction for hernia, hydrocele or phimosis.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Urine Biomarkers | 48 months
  The investigators will focus on the urine by investigating for intrarenal remodeling processes and searching for kidney-specific biomarkers by urinary single-cell and EVs screening (aim 1).
Blood Biomarkers | 48 months
  Moreover, based on the hitherto revealed capability of blood cells to perceive organ-specific illnesses, the investigators will perform WBGEP of babies with unilateral UPJO to identify early biomarkers of disease progression (aim 2).

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Univeristà degli Studi della Campania Luigi Vanvitelli, Naples, Campania
  - Department of Clinical Sciences and Community Health, University of Milano, Milan
  - Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico, Milan
  - Obstetrics and Gynecology Unit, University of Modena and Reggio Emilia, Modena
  - AORN Santobono-Pausilipon, Naples

IPD SHARING:
Plan to Share IPD: No